CLINICAL TRIAL: NCT01231932
Title: Characterizing Fatigue Experienced by Cancer Patients Receiving Primary Treatment and Cancer Survivors
Status: Terminated | Type: Observational
Why Stopped: Principal Investigator (PI) of this study is retiring.
Sponsor: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 110014; 11-NR-0014
Record Dates: First submitted 2010-10-29; First posted 2010-11-01 (Estimated); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Cancer; Fatigue; Prostate Cancer; Breast Cancer; Cancer Survivor
Keywords: Fatigue; Cytokines; Cancer Therapy; Cancer Treatment; Gene Expression Patterns; Natural History; Cancer
MeSH Terms: conditions — Neoplasms; Fatigue; Prostatic Neoplasms; Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Cancer survivors: Individuals recently completed primary treatment for cancer
- Individuals receiving cancer treatment: Individuals receiving cancer treatment
- Individuals with cancer: Individuals with cancer

SUMMARY:
Background:

- Fatigue is a common side effect of cancer and its treatment. Up to 96% of patients with cancer have fatigue. The cause of fatigue in people with cancer or those receiving treatment is poorly understood, making fatigue hard to treat. More research is necessary to understand why cancer patients experience fatigue. Previous research has shown that fatigue may be caused by a number of factors, including problems with the immune system response of the body while undergoing cancer treatment. The researchers of this study are trying to understand how the immune system and other chemicals of the body change while a person receives cancer treatment and how these changes play a role in causing fatigue. The researchers are also interested in how a person s quality of life is affected by fatigue.

Objectives:

- To study fatigue in individuals who have cancer, are receiving cancer treatment, or have completed cancer treatment.

Eligibility:

* Individuals at least 18 years of age.
* Receiving cancer treatment, OR completed primary treatment for cancer (e.g., cancer survivors), OR on active surveillance for localized cancer.

Design:

* This study involves an initial screening visit and up to three outpatient visits.
* Participants will be screened with a medical history review (can be done virtually) and blood tests. A physical exam might also occur.
* Participants undergoing cancer treatment that has a clear completion date, will have the following visits:

  * Before the start of treatment.
  * At the end of treatment.
  * At least 3 months after treatment ends.
* Participants not receiving treatment, are cancer survivors, or undergoing cancer treatment that does not have a clear completion date, will have up to 3 visits:

  * Before the start of treatment or whenever you begin the study.
  * At least 3 months after your first visit.
  * At least 3 months after your second visit.
* At each study visit, participants will complete the following tasks (some of the tasks can be done from home or virtually):

  * Questionnaires about physical activity, fatigue, depression, and quality of life (can be done at home or virtually).
  * Have blood drawn.
  * Physical activity device and journals to study how fatigue affects physical activity.
  * Optional tests:

    * Computer games testing your memory, attention, and ability to follow directions.
    * Hand grip strength test to evaluate physical strength.
* Treatment will not be provided under this study.

DETAILED DESCRIPTION:
Although the underlying mechanisms of fatigue have been studied in several disease conditions, the etiology, mechanisms, and risk factors remain elusive, and this symptom remains poorly managed at present. Longitudinal studies related to treatment-related fatigue in cancer patients have been conducted but there are limited data showing changes in molecular mechanisms before and after cancer therapy which can identify individuals who are at risk to experience fatigue during and after therapy. Fatigue is conceptualized as a multidimensional symptom which incorporates temporal, sensory, cognitive/mental, affective/emotional, behavioral, and physiological dimensions. This prospective, observational study will explore the molecular-genetic mechanisms underlying fatigue experienced by cancer patients receiving various therapies (e.g. immune therapy, hormone therapy, radiation therapy and chemotherapy).

The primary objective of the study is to describe the changes in the self-reported fatigue experienced by cancer patients over time. The secondary objectives of this study are to (1) investigate the associations between inflammatory, neurometabolic, stress, and mitochondrial markers with fatigue intensification over time during the course of treatments, (2) determine changes in gene expression from peripheral blood samples over time during the course of treatments, (3) relate changes in the levels of these biological markers (i.e., inflammatory/metabolic/stress profiles and gene expression) to patient reported outcomes (PROs) of self-reported fatigue, sleep disturbance, depression, and health-related quality of life (HRQOL) scores, (4) measure cognitive functioning, skeletal muscle strength, physical activity levels and energy expenditure of patients and relate these findings with changes in PRO scores, the inflammatory/metabolic/stress profiles and gene expression, and (5) investigate the psychometric property of the Saligan-Walitt Integrated Fatigue Tool (SWIFT).

ELIGIBILITY:
* INCLUSION CRITERIA:

To be included, patients must meet all of the following criteria:

* Medical documentation confirming diagnosis of:

  --Clinically localized or metastatic cancer as determined by diagnostic testing such as cytology and imaging (such as, but not limited to non-metastatic head and neck cancer, lung cancer, breast cancer, renal cancer); OR completed primary treatment for cancer (e.g., cancer survivors) OR on active surveillance for localized cancer;
* Able to provide written informed consent;
* Women and men greater than or equal to 18 years of age;
* NIH employees and staff are eligible to participate.

EXCLUSION CRITERIA:

* Progressive or unstable disease other than cancer of any body system causing clinically significant fatigue (e.g. class IV congestive heart failure, end-stage renal disease, stage IV chronic obstructive pulmonary disease) including patients with

  * Systemic infections (e.g., human immunodeficiency virus [HIV], active hepatitis);
  * Documented history of unstable major depression, bipolar disease, psychosis, or alcohol/drug dependence/abuse; requiring hospitalization/institutionalization;
  * Uncorrected hypothyroidism;
  * Untreated anemia;
  * Chronic inflammatory disease (e.g. rheumatoid arthritis, systemic lupus erythematosus).
* Patients regularly taking antipsychotics, and anticonvulsants, since these medications cause significant fatigue.
* NINR employees or subordinates, relatives, and/or co-workers of NINR employees/staff or study investigators.
* Self-report of color-blindness verified by taking the Ishihara card test with scores >14 (10 minutes) will be an exclusion from the Stroop Test. This card test will be administered only if the patient reports being color blind.
* Severe essential hand tremor or severe hand pain (e.g., severe arthritis or severe carpel tunnel) will be an exclusion from the computerized tests and the skeletal muscle strength test.
* Ongoing medical condition that is deemed by the Principal Investigator to interfere with the conduct or assessments of the study or safety of the participant.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study is actively enrolling patients from referrals obtained from NCI and from PRPL.
Sampling Method: Non-Probability Sample
Enrollment: 163 (Actual)
Dates: Start 2011-02-04 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2025-04-16 (Actual)

PRIMARY OUTCOMES:
Self-reported fatigue | Up to 3 times throughout study
  Self-reported fatigue

SECONDARY OUTCOMES:
The inflammatory/metabolic/stress profile; gene expression changes; self-reported fatigue; sleep disturbance; depression; HRQOL scores; cognitive function; skeletal muscle strength; physical activity levels and energy expenditure; SWIFT scores. | Up to 3 times throughout study
  The inflammatory/metabolic/stress profile; gene expression changes; self-reported fatigue; sleep disturbance; depression; HRQOL scores; cognitive function; skeletal muscle strength; physical activity levels and energy expenditure; SWIFT scores.

CONTACTS AND LOCATIONS:
Overall Officials: Leorey N Saligan, C.R.N.P., Principal Investigator — National Institute of Nursing Research (NINR)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Background] Bower JE, Ganz PA, Aziz N, Fahey JL. Fatigue and proinflammatory cytokine activity in breast cancer survivors. Psychosom Med. 2002 Jul-Aug;64(4):604-11. doi: 10.1097/00006842-200207000-00010. PMID 12140350
- [Background] Brola W, Ziomek M, Czernicki J. [Fatigue syndrome in chronic neurological disorders]. Neurol Neurochir Pol. 2007 Jul-Aug;41(4):340-9. Polish. PMID 17874343
- [Background] Miaskowski C, Paul SM, Cooper BA, Lee K, Dodd M, West C, Aouizerat BE, Swift PS, Wara W. Trajectories of fatigue in men with prostate cancer before, during, and after radiation therapy. J Pain Symptom Manage. 2008 Jun;35(6):632-43. doi: 10.1016/j.jpainsymman.2007.07.007. Epub 2008 Mar 20. PMID 18358683
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2011-NR-0014.html